CLINICAL TRIAL: NCT01061944
Title: Biopsies of Cancer Patients for Tumor Molecular Characterization
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lecia V. Sequist, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 09-369
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Cancer; Metastatic Cancer
Keywords: biopsy; tumor biopsy; genetic studies
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor biopsy
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In this research study, we are looking at performing a repeat biopsy of patients' tumors, even though they have already been diagnosed with cancer. The tumor tissue obtained from the biopsy will be studied to see what it looks like at the molecular (genetic) level. By conducting this study, we hope to learn more about how cancers work, why cancers respond to certain treatments, and how they become resistant to certain treatments. We also hope to demonstrate that biopsies like this can be performed safely in large numbers of patients. The research done on the tumor samples may help us identify which patients in the future are most likely to respond to new cancer therapies.

DETAILED DESCRIPTION:
* In order to participate in this research study, participants must have already been diagnosed with cancer. The cancer must be located in a part of the body that is accessible for a biopsy and the doctor that will perform the biopsy must agree that the participant is a good candidate for biopsy. The biopsy will be done in the usual way, as part of your standard medical care.
* After the biopsy, the participant will return to the clinic approximately one week later for a check on their status. At this visit participants will be asked questions about your post-biopsy health. We will continue to follow-up with the participants by phone or at subsequent clinic visits for one month following the biopsy.
* The biopsy obtained will be studied in the Translational Research Laboratory at Massachusetts General Hospital, where it will undergo a panel of genetic tests. These tests look to find out what is driving the cancer or making it tick. It is important to understand that the genetic tests we will do include a number of cancer related genes or proteins that may be important for making treatment decisions, either now or in the future. The test results may or may not show a finding that could affect the participant's treatment options. There will be no specific testing done for inherited genetic abnormalities, so undergoing this research will not give information about the risk of cancer for people in the participant's family.
* If there is left-over tissue from biopsy, it will also be used to try to discover new findings about how cancers respond or become resistant to cancer treatments. These experiments will include trying to grow the cancer cells in a petri dish in the lab or trying to grow the cancer cells inside research mice to learn more about how the cancer works. This portion of the testing os part of the research study and is considered experimental, so the results will not be entered into the participants' medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must already be known to have metastatic, incurable cancer.
2. Patients must have been referred for repeat tumor biopsy as part of standard care and biopsy must have been approved by the appropriate biopsy service (interventional radiology or surgery). Such approval includes review of medical history and laboratory parameters as per standard care.
3. 18 years of age or older
4. Patients must have previously responded to a molecularly-targeted therapy and subsequently developed resistance, or have an analogous clinical situation in which determining their molecular genotype is of interest clinically and/or scientifically.

No specific exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be identified by their oncologist and the service performing the biopsy as a good candidate for the repeat tumor biopsy procedure. Review of the medical record and laboratory data is also performed to ensure the risks of complications are reasonable low and within standard parameters.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2010-02; Primary Completion 2016-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and safety of repeat biopsies for molecular characterization. | 2 years

SECONDARY OUTCOMES:
To determine the somatic genotype of cancer patients with acquired resistance to a targeted therapy, and to compare these findings with pre-treatment genomic profiled from the same patients. | 2 years
To estimate the success rate of molecular diagnostics from biopsies specifically obtained for such testing. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lecia V. Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States